CLINICAL TRIAL: NCT03683186
Title: A Phase 3 Open-label Extension (OLE) Study to Evaluate the Long-term Safety and Efficacy of Ralinepag in Subjects With World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study Evaluating the Long-Term Efficacy and Safety of Ralinepag in Subjects With PAH Via an Open-Label Extension
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROR-PH-303; APD811-303 (Other: Arena Pharmaceuticals)
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: PAH; Pulmonary Hypertension; Pulmonary Arterial Hypertension; Hypertension; Connective Tissue Diseases; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Disease
Keywords: Prostacyclin; Connective Tissue Disease-Associated; 6 Minute Walk Test; 6 Minute Walk Distance; Pulmonary Vascular Resistance; Right Ventricular Function
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Hypertension; Connective Tissue Diseases; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases | interventions — ralinepag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ralinepag (Experimental): Ralinepag once daily extended-release tablets (oral) 50, 250, and 400 mcg titrated to the highest tolerated dose.
  Interventions: Drug: Ralinepag

INTERVENTIONS:
Drug: Ralinepag — Active
  Other Names: APD811

SUMMARY:
Study ROR-PH-303, ADVANCE EXTENSION, is an open-label extension (OLE) study for participants with WHO Group 1 PAH who have participated in another Phase 2 or Phase 3 study of ralinepag.

DETAILED DESCRIPTION:
Study ROR-PH-303 is a multicenter, open-label extension (OLE) study for subjects with WHO Group 1 PAH who have participated in another Phase 2 or Phase 3 study of ralinepag and who qualify for entry based upon participation in the prior study. Subjects who discontinue participation in a prior study due to safety issues related to study medication or who fail to complete study procedures will not be eligible to enter Study ROR-PH-303. Subjects who meet all OLE entry criteria will be enrolled and will receive ralinepag in addition to their pre-existing PAH disease-specific background therapy.

For subjects who are enrolled from an ongoing double-blind Phase 2 or Phase 3 ralinepag study, a 16-week blinded Dose Titration Period will be completed following enrollment into the OLE. Subjects previously on ralinepag will continue on the same dose during the Dose Titration Period as received in the original study and will also initiate placebo treatment in the OLE.

Subjects who are enrolled from a non-blinded study or another OLE will not participate in the blinded Dose Titration Period in Study ROR-PH-303 but will be enrolled directly into the Treatment Period and continue on the dose of ralinepag received in the original study.

All subjects will receive ralinepag in the OLE study until premature discontinuation of ralinepag due to an AE/serious adverse event (SAE) or other reason, marketing approval of ralinepag is granted in the region in which the study is conducted, or the study is discontinued by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study prior to initiation of any study-related procedures.
2. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Completed the protocol-defined Study Drug Termination Visit or End of Study Visit procedures in the preceding ralinepag study.
4. Both male and female subjects agree to use a medically acceptable method of contraception throughout the entire study period from informed consent through the 30 day Follow-up Visit, if the possibility of conception exists. Eligible male and female subjects must also agree not to participate in a conception process (i.e., actively attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) during the study and for 30 days after the last dose of ralinepag.

Exclusion Criteria:

1. Subjects who prematurely discontinued investigational medicinal product (IMP) due to a drug-related AE/SAE or tolerability issue in the preceding ralinepag study in which they were enrolled, or subjects who did not complete all protocol defined study procedures at a Study Drug Termination Visit or End of Study Visit in the preceding ralinepag study.
2. Subjects who withdrew consent during participation in another ralinepag study.
3. Female subjects who wish to become pregnant or who have a positive pregnancy test on Day 1 (OLE Entry Visit), or are lactating or breastfeeding.
4. Subjects who have undergone lung or heart/lung transplant or the initiation of long-term parenteral or inhaled therapy with a prostacyclin during the time since participation in their original ralinepag study.
5. Subjects who had an emergency unblinding procedure in a prior Phase 2 or 3 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events [Safety and Tolerability] | Up to 6 years
  The safety and tolerability of ralinepag will be evaluated by the Number of subjects with treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (190):
- United States (48):
  - St. Joseph's Hospital and Medical Center-Norton Thoracic Institute, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UCSD Health Sciences, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati-Medical Science Building, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - StatCare Pulmonary Consultants, Knoxville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Vermont Lung Center, Burlington, Vermont
  - Carilion Clinic Pulmonary and Sleep Medicine, Roanoke, Virginia
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (12):
  - Hospital Italiano, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital PROVINCIAL "Dr. Jose Maria Cullen", Santa Fe, Santa Fe de La Vera Cruz
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Cardiologia Palmero, Caba
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Respirar, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Instituto de Investigaciones Clinicas, Mar del Plata
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH - Elisabethinen, Fadingerstrasse 1, Linz
  - AKH Wien, Innere Med. II, Kardiologie, Währingergürtel 18-20, Vienna
- Belgium (2):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - UZ Leuven, UZ Leuven Campus Gasthuisberg, Herestraat 49, Leuven
- Brazil (7):
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia, Goiás
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Hospital Sao Lucas da PUC-RS, Porto Alegre, R.S
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP-Faculdade de Medicina da Universidade Estadual Paulista Campus Botucatu, Botucatu, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
  - Instituto do Coracao, São Paulo, São Paulo
- Bulgaria (2):
  - MHAT - "National Heart Hospital" EAD, 65, Konyovitza Str., Sofia
  - MHAT "Sveta Anna" Sofia AD, Sofia
- Canada (6):
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - LHSC - Victoria Hospital, London, Ontario
  - University Health Network-Toronto General Hospital, Toronto, Ontario
  - SMBD Jewish General Hospital d/b/a Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- Instiuto Nacional del Torax, Providencia, Santiago de Chile, Chile
- China (5):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
- Croatia (2):
  - Clinical Hospital Dubrava Zagreb, Avenija G.Šuška 6, Zagreb
  - University Clinic for Pulmonary Diseases, Jordanovac 104, Zagreb
- Vseobecna fakultni nemocnice v Praze, II. interni klinika kardiologie a angiologie VFN a 1. LF UK, U nemocnice 2, Prague, Czechia
- Denmark (2):
  - Århus Universitetshospital, Aarhus
  - Copenhagen University Hospital (Rigshospitalet), Copenhagen
- France (11):
  - CHU de Strasbourg - Nouvel Hôpital Civil, Ctre de competence Hypertension Arterielle Pulmona, 1 place de l Hopital, Strasbourg, Bas Rhin
  - CHU de Grenoble - Hôpital Albert Michallon, Clinique de Cardiologie, Boulevrad de la Chantourne, Grenoble, Isere
  - CHU Nancy - Hôpital de Brabois Adultes, Pneumologie- Oncologie Médicale, Rue du Morvan, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU de Saint-Etienne - Hopital Nord, Service de Medecine vasculaire et therapeutique, 81 Avenue A. Raimond, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Service de Pneumologie, 59 Boulevard Pinel, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Service de Pneumologie, 78 Avenue du General Leclerc, Le Kremlin-Bicêtre, Val De Marne
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHRU de Lille - Hopital Cardiologique, Lille
  - Hôpital Nord - CHU Marseille, Marseille
- Germany (8):
  - Thoraxklinik-Heidelberg Zentrum für Pulmonale Hypertonie, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitaetsmedizin der Johannes-Gutenberg-Universitaet Mainz, Zentrum für Kardiologie I, Centrum für Thrombose und Hämostase (CTH), Langenbeckstrasse 1, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum des Saarlandes, Innere Medizin V, IMED, Kirrberger Strasse 100, Gebäude 41, Homburg, Saarland
  - Universitätsklinikum Leipzig, Medizinische Klinik II, Pneumologie, Leipzig, Saxony
  - Schwarzwald-Baar Klinikum, Donaueschingen
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (4):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "Onasseio" Cardiosurgery Hospital, Hemodynamic Research and Interventional Cardiology Dept., 356, Syggrou Avenue, Athens
  - University General Hospital Attikon, Chaïdári
  - AHEPA General Hospital of Thessaloniki, A' Cardiology Clinic, 1 St. Kyriakidi Street, Thessaloniki
- Hungary (2):
  - Gottsegen György Országos Kardiovaszkuláris Intézet, Budapest
  - Pecsi Tudomanyegyetem, Szivgyogyaszati Klinika, Ifjusag u. 13., Pécs
- Israel (5):
  - The Lady Davis Carmel Medical Center, 7 Michal st., Haifa
  - Hadassah Ein Kerem Medical Center, Kiryat Hadassah, Jerusalem
  - Meir Medical Center, 59 Tshernichovski st., Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Pulmonary Institute, 39 Jabotinsky St Ground floor, Petah Tikva
  - Tel Aviv Sourasky Medical Center, 6 Weizmann St., Tel Aviv
- Italy (8):
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione (ISMETT), Palermo, PA
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, S.C. di Cardiologia, Viale Luigi Pinto, 1, Foggia
  - IRCC Ospedale Policlinico San Martino, Genova
  - Centro Cardiologico Monzino, IRCCS U.O. Scompenso, Milan
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Via Francesco Sforza 35, Milan
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Viale del Policlinico, 155, Roma
- Mexico (4):
  - CICUM San Miguel, Guadalajara, Jalisco
  - Instituto Nacional de Cardiologia Dr Ignacio Chavez Rivera, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City
  - Unidad de Investigacion Clinica en Medicina, S.C., Monterrey, N.L.
- VU Medisch Centrum, De Boelelaan 1117, Amsterdam, Netherlands
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Kardiologii z Oddzialem Intensywnego Nazdoru Kardiologicznego, M. Sklodowskiej 24a, Bialystok
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Oddział Kliniczny Chorób Serca i Naczyń z Pododdziałem Intensywnego Nadzoru Kardiologicznego, Pradnicka 80, Krakow
  - NZOZ Europejskie Centrum Zdrowia, ul. Borowa 14/18, Otwock
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Oddzial Kardiologii - F, ul. Dluga 1/2, Poznan
  - Premium Clinic Wrocław CM, Podwale 83/17, Wroclaw
- Portugal (4):
  - Hospital Garcia de Orta, E.P.E, Almada
  - Centro Hospitalar e Universitário de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. Hospital Pulido Valente, Lisbon
  - Centro Hospitalar de Santo António, E.P.E., Porto
- Romania (4):
  - Institutul de Urgenta pentru Boli Cardiovasculare "Prof. Dr. C.C. Iliescu", Sos. Fundeni nr. 258, Bucharest
  - Institutul de Pneumoftiziologie "Marius Nasta", Sos. Viilor nr. 90, Sector 5, Bucharest
  - Institutul Inimii "Niculae Stancioiu" Cluj-Napoca, Cardiologie, Str. Motilor nr. 19-21, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie "Dr. Victor Babes" Timisoara, Str. Gheorghe Adam nr. 13, Timișoara
- Serbia (3):
  - Clinical Center of Serbia, Koste Todorovica 8, Belgrade
  - Clinical Center Zemun. Clinic for internal medicine, Department of Cardiology, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Put Dr Goldmana 4, Kamenitz
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Gachon University Hospital Gil Medical Center, Incheon, Namdong-gu
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Respiratory Dept., Passeig Vall d'Hebron,119-129, Neumologia, Barcelona
  - Hospital Clinic de Barcelona, C/ Villarroel, 170, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Linköping Universitetssjukhuset, Linköping
  - Norrlands Universitetssjukhus, Hjärtcentrum, Umeå
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (7):
  - Osmangazi Uni Medical Faculty, Eskişehir, Odumpazari
  - Balcalı, Çukurova Üniversitesi Kardiyoloji ABD, Adana, Saricam
  - Mersin Üniversitesi Tip Fakültesi Ciftlikköy Kampüsü, Mersin, Yenisehir
  - Gazi University Medical Faculty Hospital, Ankara
  - Uludag Universitesi Tip Fakültesi, Gorukle Kampusu, Bursa
  - Marmara Universitesi Istanbul Pendik Egitim ve Arastirma Hastanesi, Fevzi Cakmak Mahallesi Muhsin Yazicioglu Cad. No: 10, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Mithatpasa caddesi Inciralti Balcova, Izmir
- Ukraine (3):
  - CE Dniprop RCC&C Center of Dniprop RC Dept of Card SI DMA of MOHU, Chair of Internal Medicine 3, 28, Knyazya Volodymyra Velykogo St., Dnipro
  - SI F.H.Yanovskyi National Institute of Phthisiology and Pulmonology of NAMSU, Clinical and Functional Dept, 10, Amosova St., Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Clinical Hospital, Dept of Cardiology, D.Halytskyi Lviv NMU, Ch of Internal Medicine #1, 7, Chernihivska str., Lviv
- United Kingdom (5):
  - Royal Free London NHS Foundation Trust, Pond Street, London, Greater London
  - Royal Brompton Hospital, London, Greater London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Sir William Leech Lung Research Centre, Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Golden Jubilee National Hospital, Glasgow, West Dunbartonshire
  - Hammersmith Hospital, London